CLINICAL TRIAL: NCT06660953
Title: Comparison of Intraopertaive and Postoperative Analgesic Efficacy of Ultrasound-guided Quadratus Lumborum II and Errector Spinae Plane Block in Patients Undergoing Kidney Transplantation
Brief Title: Comparison of Analgesic Efficacy ESP Block and QLB II in Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Muharrem Baturu, Asistant professor, University of Gaziantep
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ESB vs QLB in transplatation; 2022/172 (Other: University of gaziantep clinical research ethics committee)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Analgesia; Intraoperative Analgesia
Keywords: errector spina plane block; quadratus lumborum block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomised controlled clinical study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group E (Active Comparator): Group that Erector spinae plane block was applied.
  Interventions: Procedure: Erector Spinae Plane Block
- Grup Q (Active Comparator): Group that Quadratus lumborum type II block was applied
  Interventions: Procedure: Quadratus Lumborum Block (QLB)
- Group K (No Intervention): no block was applied

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — For ESP, high frequency linear ultrasound probe was planned transversely to the midline and spinous features were visualized. Cervical C7 and T7 vertebrae at the lower end of the scapula, which were accepted as landmarks, were determined and marked with a sterile surgical drawing pen. According to these landmarks, the USG probe was moved 2-3 cm laterally towards the points where kidney transplantation was planned at the T10 vertebral level, and the transverse parts, trapezius, latissimus dorsi, serratus and erector spina muscles were visualized. Using the block needle that can be visualized on USG with in-plane surgery, the skin, subcutaneous tissue and trapezius, latissimus dorsi, serratus and erector spina muscles were passed in a cranio caudal direction and the needle location was confirmed by hydrodissection with 2-5 ml of serum. The distribution of the block procedure and the spread of local anesthetic were linearly visualized with 10 ml bupivacaine and 10 ml 0.9% saline.
  Arms: Group E
Procedure: Quadratus Lumborum Block (QLB) — The QL block II was done under aseptic technique, in lateral position with the side intended to block side up. A high frequency ultrasound linear probe covered in sterile sheath was placed anterior and superior to the iliac crest. The three anterior abdominal muscles were visualized. The external oblique muscle was followed posterolaterally until its posterior border was identified. Subsequently, the probe was tilted towards the attachment site of both the internal and external oblique muscles over the quadratus (QL) muscle until the midline of the thoracolumbar fascia was seen as a bright hyperechogenic line located between the posterior border of the quadratus lumborum muscle and the middle thoraco-lumbar fascia (anterior to latissiumus dorsi and erector spinae muscles). A 22-gauge Facet-tip SonoPlex needle of appropriate length estimated from the depth and length of required needle trajectory during scout scanning was inserted via in-plane technique. The needle was directed from a
  Arms: Grup Q

SUMMARY:
Renal transplantation is an increasingly common surgery in recent years. Opioid and/or NSAID use is common in postoperative pain management. However, these drugs have many side effects. Peripheral blocks provide more effective analgesia both intra and postoperatively, and also reduce the use of systemic drugs. The aim of this study was to compare the effects of two different nerve blocks (ESP vs QLB II) on intraoperative remifentanil dose and postoperative analgesia.

DETAILED DESCRIPTION:
All patients participating in this study underwent a standard anesthesia induction and maintenance. When the patients arrived in the operating room, noninvasive blood pressure, heart rate, electrocardiogram, and oxygen saturation monitoring were performed. Intravenous administration of 2-3 mg/kg propofol, 1-2 mcg/kg Fentanyl, and 0.1 mg/kg atracurium was performed for general anesthesia induction, and then the patients were intubated. After tracheal intubation, anesthesia was maintained with 50% oxygen/air and sevoflurane. An additional 0.1 mg/kg atracurium was added during the surgery as needed. Analgesia was provided with 0.1-0.3 mcg/kg/h intravenous infusion of remifentanil, which was increased or decreased according to the patient's hemodynamics. Intravenous neostigmine was administered for neuromuscular recovery after the surgery. The patient awoke from general anesthesia. Total anesthesia duration, hemodynamic data, and remifentanil dose were recorded.

Patients who would receive a block after general anesthesia induction were randomly determined. These patients were placed in the lateral decubitus position and ESP block or QLB II was applied under ultrasound guidance and echogenic needle (Techniplex 18 gauge; 100 mm needle, Vygon value life) under aseptic conditions. All interventions were performed by an experienced anesthesiology specialist. All procedures were performed under ultrasound guidance using a linear probe (Logiq e GE 12L-RS linear probe, GE LOGIQ e Ultrason device). Patients were randomly divided into 3 groups. Patients who underwent ESB were named Group E, those who underwent QLB were named Group Q, and patients who did not receive a block were named the control group.

The QL block II was done under aseptic technique, in lateral position with the side intended to block side up. A high frequency ultrasound linear probe covered in sterile sheath was placed anterior and superior to the iliac crest. The three anterior abdominal muscles were visualized. The external oblique muscle was followed posterolaterally until its posterior border was identified. Subsequently, the probe was tilted towards the attachment site of both the internal and external oblique muscles over the quadratus (QL) muscle until the midline of the thoracolumbar fascia was seen as a bright hyperechogenic line located between the posterior border of the quadratus lumborum muscle and the middle thoraco-lumbar fascia (anterior to latissiumus dorsi and erector spinae muscles). A 22-gauge Facet-tip SonoPlex needle of appropriate length estimated from the depth and length of required needle trajectory during scout scanning was inserted via in-plane technique. The needle was directed from anterolateral to posteromedial after making a negative aspiration test with aliquots of 0.5 ml saline to confirm hydrodissection in the lumbar interfascial triangle (LIFT) between the QL muscle and middle thoracolumbar fascia. An injection of LA was given according to the group allocated. Aliquots of LA with intermittent aspiration during injection was performed in the desired confirmed space After the needle tip was correctly positioned, 10 ml of bupivacaine and 10 ml of 0.9% saline solution were injected.

For ESP, high frequency linear ultrasound probe was planned transversely to the midline and spinous features were visualized. Cervical C7 and T7 vertebrae at the lower end of the scapula, which were accepted as landmarks, were determined and marked with a sterile surgical drawing pen. According to these landmarks, the USG probe was moved 2-3 cm laterally towards the points where kidney transplantation was planned at the T10 vertebral level, and the transverse parts, trapezius, latissimus dorsi, serratus and erector spina muscles were visualized. Using the block needle that can be visualized on USG with in-plane surgery, the skin, subcutaneous tissue and trapezius, latissimus dorsi, serratus and erector spina muscles were passed in a cranio caudal direction and the needle location was confirmed by hydrodissection with 2-5 ml of serum. The distribution of the block procedure and the spread of local anesthetic were linearly visualized with 10 ml bupivacaine and 10 ml 0.9% saline.

The control group received 0.1 mg/kg morphine subcutaneously 30 minutes before the end of the operation. All patients were connected to a patient-controlled analgesia device (1 mg Fentanyl/100 ml saline, 2 ml bolus dose, 15 min lock, infusion rate 2 ml/h).

Postoperatively, total 24-hour fentanyl consumption and pain scores of all patients were recorded according to the visual analog scale at 1, 2, 3, 4, 6, 12 and 24 hours.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Patients with a history of allergy to general and local anesthetics to be used, inability to understand or participate in pain scoring, inability to use the PCA pump, or conditions that prevent the performance of trunkal blocks (anatomical or postoperative deformations in the region)

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of postoperative analgesia | postoperative 24 hours
  visuel analog score < 3

SECONDARY OUTCOMES:
consumption of add analgesic dos | postoperative 24 hours
  Reduction in consumption of additional analgesic administered (fentanyl PCA)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Atici E, Arslan ZI, Yilmaz H. Effect of erector spinae plane block on postoperative intravenous morphine consumption in open subcostal nephrectomy: A prospective randomized clinical trial. Agri. 2024 Jan;36(1):13-21. doi: 10.14744/agri.2022.71602. PMID 38239121
- [Result] Kolacz M, Mieszkowski M, Janiak M, Zagorski K, Byszewska B, Weryk-Dysko M, Onichimowski D, Trzebicki J. Transversus abdominis plane block versus quadratus lumborum block type 2 for analgesia in renal transplantation: A randomised trial. Eur J Anaesthesiol. 2020 Sep;37(9):773-789. doi: 10.1097/EJA.0000000000001193. PMID 32175985
- [Result] Kim Y, Kim JT, Yang SM, Kim WH, Han A, Ha J, Min S, Park SK. Anterior quadratus lumborum block for analgesia after living-donor renal transplantation: a double-blinded randomized controlled trial. Reg Anesth Pain Med. 2024 Aug 5;49(8):550-557. doi: 10.1136/rapm-2023-104788. PMID 37704438
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/37971133/